CLINICAL TRIAL: NCT06220032
Title: ANTICIPATE: Prevention of ANThracycline-Induced Cardiac Dysfunction by Dexrazoxane In PATients With diffusE Large B-cell Lymphoma: a Phase III National Multicenter Prospective Randomized Open-label Trial
Brief Title: Prevention of Anthracycline-Induced Cardiac Dysfunction With Dexrazoxane in Patients With Diffuse Large-B Cell Lymphoma
Acronym: HO170DLBCL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: UMC Utrecht (Other); Amsterdam University Medical Centers (Unknown); The Dutch Network for Cardiovascular Research (WCN) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HO170 DLBCL-ANTICIPATE; 2023-505377-32 (Other: EU CT number)
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-10

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
Keywords: dexrazoxane; primary prevention; cardiotoxicity; heart failure; diffuse large B-cell lymphoma; R-CHOP; FL; R2CHOP; LVEF
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Cardiotoxicity; Heart Failure; Lymphoma, Large B-Cell, Diffuse | interventions — Dexrazoxane; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; Lenalidomide; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Standard R-CHOP 21 treatment regimen:
  6 cycles R-CHOP 21 (rituximab*, cyclophosphamide, doxorubicin, vincristine, prednisolone)
  *The use of a biosimilar is allowed.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone; Drug: Lenalidomide; Drug: Pegfilgrastim
- Arm B - (Experimental): Addition of the cardioprotectant dexrazoxane to the R-CHOP 21 regimen:
  R-CHOP21 (rituximab*, cyclophosphamide, doxorubicin, vincristine, prednisolone plus dexrazoxane).
  *The use of a biosimilar is allowed.
  Interventions: Drug: Dexrazoxane; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone; Drug: Lenalidomide; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Dexrazoxane — Day 1 Cycle 1-6: Dexrazoxane 500 mg/m2 (iv) will be given 30 minutes before doxorubicin infusion and should be infused during 15 minutes.
  Other Names: Cardioxane
  Arms: Arm B -
Drug: Rituximab — Day 1 Cycle 1-6: 375 mg/m2 (iv)
Drug: Cyclophosphamide — Day 1 Cycle 1-6: 750 mg/m2 (iv)
Drug: Doxorubicin — Day 1 Cycle 1-6: 50 mg/m2 (iv)
Drug: Vincristine — Day 1 Cycle 1-6: 1.4 mg/m2 (max 2 mg) (iv)
Drug: Prednisolone — Day 1-5 Cycle 1-6: 100 mg (oral)
Drug: Lenalidomide — Day 1-14 Cycle 1-6: 15 mg day (oral) Only in case of a double hit lymphoma.
  Other Names: Revlimid
Drug: Pegfilgrastim — 6 mg (1 dose per cycle) in case of neutropenia. Pegfilgastim is mandatory in patients that receive R2-CHOP21.
  Other Names: Pegfilgastim

SUMMARY:
Patients treated for DLBCL are at high risk of developing AICD. This adverse event is characterized by irreversible damage to the heart muscle with a loss of cardiomyocytes and subsequent decline in cardiac pumping capacity. Thereby patients treated for this malignancy are at double the risk of developing symptomatic heart failure / cardiomyopathy when compared to the general population. This corresponds to a cumulative incidence of 5-10% within 5-years after receiving R-CHOP. In the elderly, an incidence of 26% has been reported after 8-years of follow-up. Among patients who die in complete remission, heart failure has been described to be one of the most important causes of death. ANTICIPATE aims to evaluate if dexrazoxane can prevent AICD in DLBCL patients and identify those at highest risk of AICD. Of all patients treated with anthracyclines in a first-line setting, DLBCL patients were chosen for this trial for two primary reasons. Firstly, these patients have a favourable oncological prognosis with a 5-year relative survival in the Netherlands of 64-78% in those aged 18-74 years increasing the importance of preventing long-term toxicity. Secondly, the cumulative anthracycline dose used for the treatment of DLBCL is higher than the dose used in breast cancer. The cumulative anthracycline dose is the most important risk factor for AICD known.

DETAILED DESCRIPTION:
HO170 DLBCL-ANTICIPATE: "Prevention of ANThracycline-Induced Cardiac dysfunction by dexrazoxane In PATients with diffusE large B-cell lymphoma" is a national randomized controlled trial that will be conducted across 25 Dutch hospitals. This study will include adult patients with DLBCL in which first-line treatment with 6 cycles of R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) is planned (cumulative doxorubicin dose 300 mg/m2). In this trial, we have chosen to include patients with a normal cardiac function before chemotherapy because cardiac dysfunction is a contra-indication for administration of anthracyclines. A total of 324 DLBCL patients will prior to treatment be randomized in a 1:1 ratio to either (1) intravenous dexrazoxane administration in a 10:1 dexrazoxane:doxorubicin ratio prior to each doxorubicin infusion or (2) no cardioprotective treatment (current standard of care). Due to the low pH of the dexrazoxane solution that would jeopardize the blinding no placebo is used. Cardiac function will be screened with echocardiography prior to the initiation of chemotherapy and followed-up at 4- and 12-months post randomization. The primary end point of the study will be the incidence of AICD, defined as a left ventricular ejection fraction (LVEF) decline of ≥10 percentage points from baseline and below 50% (normal reference value for two-dimensional (2D) echocardiography). The secondary endpoint will be the percentage of patients with complete metabolic remission (CMR) after R-CHOP chemotherapy, to reassure that dexrazoxane does not influence the antineoplastic efficacy of doxorubicin. To declare ANTICIPATE successful, the trial must show both the superiority of addition of dexrazoxane on the primary endpoint and non-inferiority on the secondary endpoint. Deep-phenotyping of patient- and treatment-related factors will be performed to evaluate their prognostic value.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated patients with a confirmed histologic diagnosis of CD20+ DLBCL according to WHO classification 2022:

   * DLBCL, not otherwise specified (NOS)
   * High-grade B-cell lymphoma NOS
   * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 translocation when DA-EPOCH-R is not an option. R2- CHOP is allowed.
   * Follicular lymphoma
   * T-cell/histiocyte-rich B cell lymphoma (THRBCL)

   Note: Transformed, previously untreated lymphoma is allowed.

   Note: 5-day treatment of dexamethasone 15 mg/day or prednisone 100 mg/day or local radiotherapy in order to control life-threatening/invalidating tumor related symptoms is allowed.

   Note: It is allowed to start with a first cycle of R-CHOP21 pending the FISH results.
2. Planned treatment with 6 R-CHOP21. The following regimens are also allowed:

   * Treatment with reversed R-CHOP21
   * Treatment with R2-CHOP21 (6 R-CHOP21 + lenalidomide 15 mg day 1-14) in case of double hit lymphoma
   * Two additional administrations of rituximab after 6 cycles of R-CHOP21
   * High dosis MTX and/or MTX-it for CNS prophylaxis
3. Ann Abor stages II-IV and stage I if the treatment plan is 6 R-CHOP21 in case of bulky disease (defined as a ≥10 cm mass);
4. Age ≥ 18 years;
5. WHO performance status ≤ 2, WHO 3 performance status is allowed when considered directly related to the DLBCL;
6. Negative pregnancy test at study entry for women of childbearing potential;
7. Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agrees to practice two effective methods of contraception, at the same time, from the time of signing the informed consent through at least 12 months after the last dose of protocol treatment, or agrees to completely abstain from heterosexual intercourse;
8. Male patient, even if surgically sterilized, (i.e., status post vasectomy) agrees to practice effective barrier contraception during the entire study period and through 12 months after the last dose of protocol treatment, or agrees to completely abstain from heterosexual intercourse;
9. Patient is able to adhere to the study visit schedule and other protocol requirements;
10. Written informed consent.

Exclusion Criteria:

1. Any of the following B-cell lymphomas according to WHO classification 2022:

   o Central Nervous System involvement by DLBCL;

   Note: high CNS-IPI is allowed
   * Testicular DLBCL;
   * Primary mediastinal B-cell lymphoma;
   * Epstein-Barr virus (EBV) post-transplant lymphoproliferative disorder;
2. Any prior malignancy or present malignancy other than DLBCL that required or requires systemic therapy. Prior surgery or local radiotherapy is allowed in case the heart has not been exposed.
3. Patients requiring treatment with mini-R-CHOP
4. Pre-existing cardiac disease including:

   * LVEF <50% measured with echocardiography (2D or 3D)
   * Symptomatic heart failure (NYHA ≥II) or hospitalization for heart failure in the last year;
   * Refractory anginal symptoms
   * Cardiac arrhythmias not controlled with optimal medical treatment, in case of atrial fibrillation the ventricular response needs to be <110/min;
   * Significant valvular dysfunction on echocardiography;
   * Non-ischemic cardiomyopathy
5. Non-diagnostic/poor transthoracic echocardiography imaging quality at baseline;
6. Severe pulmonary dysfunction defined as breathlessness at rest (COPD GOLD III or IV), unless clearly related to DLBCL;
7. Severe neurological or psychiatric disease;
8. Inadequate hematological function (absolute Neutrophil Count (ANC) <1.0x109/L or platelets <75x109/L), unless clearly related to DLBCL;
9. Significant hepatic dysfunction (serum bilirubin or transaminases ≥ 3 times the upper limit of normal) unless related to lymphoma infiltration of the liver;
10. Active hepatitis B or C infection (serology testing is required at screening). Patients positive for hepatitis B surface antigen (HBsAg) regardless of antibody status or HBsAg negative but anti-HBc positive are only eligible if HBV-PCR is negative and patients are protected with lamuvidine or entecavir. Patients with positive hepatitis C serology are only eligible if HCV-(RNA) is confirmed negative;
11. Significant renal dysfunction (creatinine clearance < 30 ml/min after rehydration) or requiring dialysis;
12. Active uncontrolled fungal, bacterial and/or viral infection;
13. Patient known to be HIV-positive;
14. Breast-feeding female patients;
15. Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule;
16. Participation in another clinical trial with anti-cancer therapy or a cardiovascular drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of AICD. | 12 months after LPI
  The incidence of AICD (measured with 2D) within 12 months after registration.

SECONDARY OUTCOMES:
Complete Metabolic Remission. | 12 months after LPI
  Complete metabolic remission (CMR) on 18F-FDG PET-CT at end of treatment 6-8 weeks after completion of 6x R-CHOP21.
Overall survival (OS). | 12 months after LPI
  Overall survival (OS) at 12-months.
Progression-free survival. | 12 months after LPI
  Progression-free survival (PFS) at 12-months.
LVEF and global longitudinal strain (GLS). | 12 months after LPI
  LVEF (2D and 3D) and global longitudinal strain (GLS) at end of treatment and 12-months after start of treatment.
NYHA. | 12 months after LPI
  NYHA functional class.
Cardiac biomarkers. | 12 months after LPI
  Release of cardiac biomarkers. At entry, after every cyle of R-CHOP, at EOT and FU. CK (if available); CK-MB (if available) & (hs)Troponin T/I (assay according to local practice).
Quality of Life. | 12 months after LPI
  To analyse the impact of the addition of dexrazoxane on QoL via validated questionaires such as QLQ-C30, NHL-HG29, PRO-CTCAE.

OTHER OUTCOMES:
Safety and toxicity. | 12 months after LPI
  Safety and toxicity as defined by type, frequency and severity of adverse events as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Secondary malignancies. | 12 months after LPI
  Incidence of secondary malignancies.
Major Adverse Cardiovascular Events. | 1- 2-, 5- and 10 years
  Major Adverse Cardiovascular Events (MACE) at 1-, 2-, 5- and 10-years.

CONTACTS AND LOCATIONS:
Overall Officials: A. van Rhenen, MD, Principal Investigator — UMC Utrecht; M.P.M. Linschoten, MD, Principal Investigator — Amsterdam UMC
Locations (25):
- Netherlands (25):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Almelo-ZGTALMELO, Almelo
  - NL-Amstelveen-AMSTELLAND, Amstelveen
  - NL-Apeldoorn-GELREAPELDOORN, Apeldoorn
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Breda-AMPHIA, Breda
  - NL-Delft-RDGG, Delft
  - NL-Dordrecht-ASZ, Dordrecht
  - NL-Eindhoven-CATHARINA, Eindhoven
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Goes-ADRZ, Goes
  - NL-Groningen-MARTINI, Groningen
  - NL-Harderwijk-STJANSDALHARDERWIJK, Harderwijk
  - NL-Hilversum-TERGOOI, Hilversum
  - NL-Hoofddorp-SPAARNEGASTHUIS, Hoofddorp
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Nijmegen-CWZ, Nijmegen
  - NL-Rotterdam-IKAZIA, Rotterdam
  - NL-Schiedam-FRANCISCUSVLIETLAND, Schiedam
  - NL-Sittard-ZUYDERLAND MC, Sittard
  - NL-Sneek-ANTONIUSSNEEK, Sneek
  - NL-Den Haag-HAGA, The Hague
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Venlo-VIECURI, Venlo
  - NL-Zwolle-ISALA, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
According to the current publication policy the protocol and Statistical Analysis Plan (SAP) will be shared. The Principal Investigators can be contacted for IPD sharing after the publication of the study results. According to the 'HOVON Sample and/or Data request Form' the HOVON director; chair of the lymphoma working group, the study PI and Coordinating Investigator should approve data/sample sharing.
Supporting Information: Study Protocol, SAP
Time Frame: After the publication of primary endpoint analysis.

REFERENCES:
- [Derived] Linschoten M, Geels J, van Werkhoven E, Visser-Wisselaar H, Chamuleau MED, Teske AJ, Robbers L, Oerlemans S, Crommelin H, Breems-de Ridder M, Schut A, Asselbergs FW, van Rhenen A; HOVON 170 DLBCL - ANTICIPATE consortium. Rationale and design of the HOVON 170 DLBCL-ANTICIPATE trial: preventing anthracycline-induced cardiac dysfunction with dexrazoxane. Cardiooncology. 2025 Jan 28;11(1):8. doi: 10.1186/s40959-025-00303-y. PMID 39875951
- See also: HOVON study website — https://hovon.nl/nl/trials/ho170